CLINICAL TRIAL: NCT02694510
Title: Impact of Protecting TPN Solution From Light on the Oxidant-antioxidant State of Preterm Infant
Brief Title: Light Protection of TPN and Oxidative Stress in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Assistant professor, PhD, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MS/299
Record Dates: First submitted 2016-02-16; First posted 2016-02-29 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Oxidative Stress in Preterm Infants
Keywords: Preterm infants; Oxidative stress; Parenteral nutrition
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Light-protection (Active Comparator): Light-protection of TPN solutions. TPN bags and infusion sets will be protected from light by aluminum foils throughout the study period.
  Interventions: Other: Light-protection of TPN solutions
- Light-exposure (Active Comparator): TPN bags and infusion sets will be exposed to light throughout the study period.
  Interventions: Other: Light-protection of TPN solutions

INTERVENTIONS:
Other: Light-protection of TPN solutions — TPN bags and infusion sets in the Light-protected group will be covered by aluminum foils to protect the inside TPN solution from exposure to ambient or photo-therapy lights in the NICU. Protection will be made throughout the study period until the infant reaches full feeding and TPN is discontinued.

SUMMARY:
Urinary peroxides and plasma glutathione/glutathione disulfide (GSH/GSSG) ratio will be measured in preterm infants less than 32 weeks gestation before and 7 days after receiving either Light-protected (Group 1) or Light-exposed (Group 2) Total Parenteral Nutrition (TPN) solutions.

DETAILED DESCRIPTION:
This study will be a prospective single blinded randomized control trial.

Inborn preterm infant less than 32 wks gestational age, receiving TPN in neonatal intensive care unit (NICU) of Mansoura University Children's Hospital as a part of their care will be included.

Preterm infant will be randomly divided into 2group:- Group 1 includes preterm infant who will receive their TPN through bags and tubing system that are protected from light by aluminum foil.

Group 2 includes preterm infant who will receive their TPN through bags and tubing system that are exposed to light.

Randomization will be done using random table technique with opaque sealed envelopes containing the serial number and the group to which the subject will be enrolled.

These envelopes will be kept in the unit ready for use at any time; each one has a number which is the serial number of the baby and group of TPN to which the baby will be enrolled.

The urine sample will be sent to the laboratory with this serial number with no information about the group of study to which this sample follows for peroxide level as well as blood sample for GSH\GSSG.

Two blood samples and two urine samples will be collected. The first one will be at 0 hour before starting TPN regimen as a base line and the second will be at 7 days of starting TPN regimen. Blood sample will be at least 1cc of blood for GSH/GSSG assay. Urine collection bag will be placed on the infant to obtain minimum of 1cc of urine for urinary peroxide level assay.

Other secondary outcomes will be assessed with duration of NICU admission including death and /or bronchopulmonary dysplasia in preterm infant at time of hospital discharge, necrotizing enterocolitis (NEC), sepsis with positive blood cultures, length of hospital stay, retinopathy of prematurity (ROP), time to full enteral feeding, duration of respiratory support, liver function, cholestasis defined as an elevated serum conjugated bilirubin >2 mg/dL, and metabolic response.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant less than 32 weeks gestational age

Exclusion Criteria:

* Infant with major congenital anomalies
* Infant of diabetic or hypertensive mother

Ages: 24 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Oxidant-antioxidant state | 7 days
  Measurement of urinary peroxides and serum GSH/GSSG ratio

SECONDARY OUTCOMES:
Death and/or Bronchopulmonary dysplasia | 60 days
  Death before hospital discharge and/or development of Bronchopulmonary dysplasia defined as oxygen requirement more than 30% fraction of inspired oxygen (FIO2) by 36 weeks corrected gestational age
Necrotizing enterocolitis as Bell's stage 2 or more | 60 days
  Necrotizing enterocolitis defined by the modified by Bell's staging criteria
Sepsis | 60 dyas
  clinical signs of sepsis confirmed by positive blood culture
Retinopathy of prematurity pre-threshold and threshold stages | 60 dyas
  Pre-threshold and threshold stages of retinopathy of prematurity will be assessed as per our NICU routine by ophthalmology specialist.
Time to full feeding | 30 days
  Time required to reach full enteral feeding and discontinue TPN
Duration of respiratory support | 60 days
  Duration of mechanical ventilation, non-invasive ventilation, and oxygen therapy
Neonatal cholestasis | 60 days
  Defined as an elevated serum conjugated bilirubin >2 mg/dL (34.2 micromoles/ l)
Metabolic disturbance | 60 days
  Episodes of hypoglycemia less than 60 mmol/L, metabolic acidosis with pH less than 7.25 and base deficit more than 10 milliequivalent/L
Length of hospital stay | 60 days
  Duration of admission to the neonatal care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, El Dakahlya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided